CLINICAL TRIAL: NCT04985461
Title: Minimally Invasive Dental Occlusion Ties Clinical Trial
Brief Title: Minimally Invasive Dental Occlusion Ties
Status: Completed | Type: Observational
Sponsor: Altru Health System (Other)
Responsible Party: Principal Investigator, Alan Johnson, Chair of Otolaryngology, Principal Investigator, Altru Health System
Other Study IDs: ENT-002
Record Dates: First submitted 2021-06-22; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Jaw Fractures; Jaw; Fracture, Upper Jaw; Mandibular Fractures; Maxilla Fracture; Jaw Fixation
Keywords: jaw fractures; mandibular fractures; maxilla fracture; jaw fixation; maxillo-mandibular fixation
MeSH Terms: conditions — Jaw Fractures; Maxillary Fractures; Mandibular Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: dental occlusion ties maxillo-mandibular fixation — This research study is being done to determine if dental occlusion ties can adequately align and stabilize jaw fractures. The chief goal of jaw fracture repair is to ensure that the teeth align normally. Traditionally, alignment has been accomplished by using steel wires and bars ("having the jaw wired"). Dental occlusion ties are newer devices similar to cable ties or "zip ties" that are wrapped around and/or between some of the teeth and secured. This procedure is intended to hold the teeth in similar alignment as wires, yet with less application time and less damage to the gums.
  Other Names: maxillo-mandibular fixation

SUMMARY:
Patients sustaining fractures of the upper (maxilla) and/or lower (mandible) jaw may be candidates for the minimally invasive technology evaluated in this study. Patients will be offered standard care including steel jaw wires or the polymer-based "zip tie"-like devices to be studied. Written consent with a full explanation of traditional "jaw wiring" techniques versus this experimental approach will be obtained from the patient. As mandible and maxilla fractures are typically treated under general anesthesia in the operating room, the devices will be applied to the patient's dentition while under general anesthetic. An exception to this will be minimally displaced or easily reduced fractures that can be treated by applying these devices in clinic under topical or local anesthetic. (Of note, wire-based techniques have been used for decades in a clinic-based application for such minimally or easily-reduced fractures.) The devices will allow stabilizing forces to the dental occlusion, achieving a similar function to temporary steel wire techniques ("arch bars"). This will allow the surgeon/principal investigator to treat the fractures with standard techniques such as applying titanium plates applied to the bone with titanium screws (known as "open reduction with internal fixation") or with sustained immobilization for 1-6 weeks (known as "closed reduction"). Note the devices are approved for 3 weeks duration. If treatment requires more than 3 weeks of immobilization, the devices will be removed and new devices re-applied. The experimental devices will be used solely as a replacement for wire-based techniques to achieve an immobile, stable jaw. If for any reason the required forces needed for jaw fracture stabilization are deemed inadequate with the experimental devices, standard steel wire techniques will be employed.

DETAILED DESCRIPTION:
Background: Mandible fractures are the second most common facial fractures behind nasal fractures. Like other fractures in the body, immobilization of the fractured segments is required for healing. For various fractures, immobilization can be achieved through casts, surgically-implanted hardware (plates, rods, screws), and other methods. Jaw fractures (mandible and maxilla) benefit from their unique connection to dentition. As the teeth are rigidly connected to the mandible and maxilla, jaw fractures can be immobilized by immobilizing the teeth in anatomic orientation. Placing the teeth in anatomic orientation (known as "dental occlusion") ensures that the cusps and the facets of the teeth fit appropriately as the fracture heals. The process of achieving this positioning is referred to as maxillo-mandibular fixation. The current leading technology to achieve maxillo-mandibular fixation (MMF) is "jaw wiring," commonly referred to as "arch bars" by facial trauma surgeons. Arch bars have been a standard of care for decades and almost invariably require application under general anesthetic for patient tolerance. Alternative variations of jaw wiring include Ivy loops, Ernst ligatures, and screw fixation approaches - all of which have achieved minimal adoption because of significant drawbacks. Wire-based MMF techniques commonly use 24 gauge stainless steel wires. The alternative wiring techniques (i.e., Ivy loops, Ernst ligatures) offer speed of application, but still require considerable manipulation by the surgeon in an operating room to apply them to the patient. The screw fixation techniques pose risks to tooth roots and to the gingiva (gums) and have also shown very limited clinician adoption.

All of these techniques, including the more widely adopted arch bars, induce considerable trauma to the gums and mucosa of the patient, causing considerable pain. Also, as these techniques are applied in the operating room under general anesthesia, the techniques incur considerable cost due to the time-consuming nature of these techniques. Further, the metal wires used in these techniques can be rigid and pointed, placing the surgical team at risk for sharps injuries.

Thus, there is a need for improved devices, systems and methods for achieving maxillo-mandibular fixation in a manner that can minimize patient discomfort, avoid the intensive labor and financial demands of such approaches, and provide a safer application for the surgical team.

This observational clinical trial aims to assess the 1) efficacy of treating mandible/maxilla fractures, 2) efficiency of application, 3) tissue trauma characteristics of a novel new cable tie-like device system used to replace wire-based techniques of maxillo-mandibular fixation, 4) the potential for these devices to be successfully applied in a clinic setting, 5) the post-treatment course for patients treated with prolonged stabilization (typically 1-6 weeks of maxillo-mandibular fixation), 6) patient's experience while wearing dental occlusion ties, and 7) the surgeon's experience with and impression of these new devices.

Study Design:

This study is a prospective, non-controlled clinical trial designed to obtain initial clinical data to further establish:

1. the clinical indications for the technology
2. appropriate sites of application for the technology (operating room and/or clinical setting)
3. clinician and patient experience during application and treatment with the devices, and
4. initial outcomes data.

Objective data such as operating room times, fracture patterns, and length of treatment will be recorded on three study forms (1. Treatment application data collection form, 2. Patient data collection form, and 3. Post-treatment data collection form). These forms also solicit subjective, unprompted data that can assist in collecting insights from the patients and the study surgeons that may not otherwise have been anticipated. Prior experiments including bench testing, cadaver testing, and a small feasibility trial have been completed in anticipation of this study.

Human subject participation:

Human subjects will be recruited through already existing referral patterns for patient care. Patients sustaining mandible or maxilla fractures and seeking care at Altru Health System may participate.

Inclusion criteria include: patients sustaining any form of mandible or maxilla fracture.

Exclusion criteria include:

1. patients with inadequate dentition (ie an edentulous patient),
2. patients under 12 years of age,
3. patients with comminuted mandible and/or maxilla fractures requiring advanced trauma techniques,
4. patients unable to consent due to intoxication, mental illness, or unconscious state, and
5. patients who are pregnant.

Data collection:

Data will be collected from the treating surgeon using the Treatment Application Data Collection Form and the Post-treatment Data Collection Form. Data will be collected from the patient using the Patient Data Collection Form. These three forms are intended to be a concise way to obtain specific data and sentiments about the patient's and surgeon's experience with the device/system. Additional data such as CT scan information will be obtained from the patient's medical record.

The output of this study will be a prospective case series manuscript describing the use of minimally invasive maxillo-mandibular fixation ties. As such, standard clinical data such as CT reports, clinical histories, and operating room times will be assessed and described in the future manuscript. This data will be stored in the standard clinical electronic medical record (EPIC). The patient's electronic medical records will be accessed subsequently for data compilation, but when this data is obtained any PHI will be immediately de-identified and linked to a patient-specific letter code (for example, patient A). The de-coding list will be kept as a hard copy stored in a physically locked cabinet in the principal investigator's office. Any paper ("hard copy") data will have the patient's name and other identifiable data replaced with this unique letter-specific identifier. All hard copy data will be shredded at the end of the study. All pictures will be electronically stored in the patient's electronic medical record, through standard electronic medical record and operating room processes. Photographs, CT images, and other electronic files (ie an MRI image) for future manuscript and presentation publication will be stored on a single password-protected USB "thumb" drive in the locked cabinet. Any pictures used in future manuscripts or presentations or posters will show patient dentition but a minimal view of the patient's face - for example approximately the lower one third of the face. This could include the upper aspects of the chin and of the nostrils of the nose, but no other anatomic features beyond these anatomic landmarks. Patients will have consented to this level of photography prior to any involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients sustaining any form of mandible or maxilla fracture

Exclusion Criteria:

* Patients with inadequate dentition (ie an edentulous patient)
* Patients under 12 years of age
* patients with comminuted mandible and/or maxilla fractures requiring advanced trauma techniques
* patients unable to consent for him/herself due to intoxication, mental illness, or unconscious state, and
* patients who are pregnant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in this study are those with mandible and/or maxilla fractures treated at a level II trauma hospital in a rural U.S. setting.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
fracture reduction | typically within the first 24 hours after surgery
  Patients will be assessed after treatment with a CT scan to assess if the fracture has been reduced or not (This is a binary variable as stated by the radiologist reading the study).
fracture healing | 6 weeks post-operatively
  Patients will be evaluated in clinic for post-operative healing. Those discharged from clinic without a need for hardware removal or revision surgery will be considered healed. (This is a binary variable - healed vs not-healed.)

SECONDARY OUTCOMES:
efficiency of application - number of ties applied | intra-operative or immediately post-operative
  The number of dental occlusion ties applied will be recorded on the surgeon post-operative data collection form.
efficiency of application - time required for surgery | intra-operative or immediately post-operative
  The operative time recorded in minutes from case start to case end.

CONTACTS AND LOCATIONS:
Locations (1):
- Altru Health System, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No